CLINICAL TRIAL: NCT05774613
Title: Bioavailability of Antioxidant Compounds and Effect on Markers of Inflammation by Ingestion of a Hibiscus Sabdariffa Beverage With Glicemic and Insulinemic Response
Brief Title: Effect of Hibiscus Sabdariffa Beverage
Acronym: Hibiscus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Tecnológico y de Estudios Superiores de Occidente (Other)
Collaborators: Instituto Tecnológico de Tepic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Hibiscus Sabdariffa
Record Dates: First submitted 2023-01-12; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Markers of Inflammation; Hyperglycemia, Postprandial; Hyperinsulinism
Keywords: Immunomodulator; Hypoglycemic; Inflammation; Post-prandial reponse; Glycemic Regulation
MeSH Terms: conditions — Hyperglycemia; Hyperinsulinism; Inflammation

STUDY DESIGN:
Intervention Model Description: Clinical trial in which both treatments under study (experimental and control) are administered to each patient at successive administered to each patient in successive periods that have been randomly determined, allowing each subject to be his or her own control. Randomly determined, allowing each subject to be his or her own control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): beverage with physical and sensory characteristics to the treatment beverage without the bioactive compounds corresponding to the study.
  Interventions: Dietary Supplement: Effect of a Hibiscus sabdariffa beverage
- Hibiscus-based drink (Experimental): beverage in patent process with application number MX/a/2022/010704
  Interventions: Dietary Supplement: Effect of a Hibiscus sabdariffa beverage

INTERVENTIONS:
Dietary Supplement: Effect of a Hibiscus sabdariffa beverage — Hibiscus sabdariffa concentrate 60 mL from improved Mexican variety , administered on a single occasion

SUMMARY:
There are numerous plant foods that are a source of bioactive compounds, which can induce an anti-inflammatory effect on various pathways of inflammatory processes in the body as it may be useful in decreasing markers of inflammation expressed by COVID-19 infectious disease and conditions such as obesity and its comorbidities. Given the above, Hibiscus sabdariffa hibiscus possesses advantages as a potential adjuvant in the management of COVID-19, as studies on the phytochemical properties of H. sabdariffa show that it has several health benefits, and could be used as a potent material for the therapeutic treatment of various diseases. Due to its high content of bioactive compounds, these can exert antioxidant, anti-inflammatory and anticarcinogenic effects, as well as help control blood glucose levels, prevent cardiovascular disease and obesity. In addition, it is a traditional component of the Mexican diet, of common consumption, easy incorporation in the diet, versatility in preparation and national production.

Therefore, to evaluate the bioavailability of bioactive compounds present in a beverage developed from the TECNM/ITESO collaboration, as well as the glycemic and insulinemic response produced by its consumption; besides establishing the effect on some inflammation markers that may be activated as a consequence of the SARS-COV-2 virus infection. This will help to increase knowledge about potential treatment/prevention schemes, avoid the development of severe manifestations of the disease, as well as boost the production and market of a national product.

DETAILED DESCRIPTION:
The following study will be carried out in two stages where an acute single-blind, crossover, randomized, single-blind clinical study will be performed, where 12 volunteers between 18 and 40 years of age, normal weight (BMI 18.5-24.9 kg/m2), without existing pathologies and/or with pharmacological treatment will be required. The characteristics of the study will be explained to the volunteers beforehand, and those who agree with the specifications will sign the informed consent form and become candidates to participate. The study will consist of the administration of a treatment drink based on hibiscus (H. sabdariffa), controlled with a placebo drink, both with a volume of 60 ml.

The first stage will consist of the selection of volunteers who will undergo two interventions. On the day of the 1st intervention, participants will arrive at 7 a.m., central time in Mexico, with an overnight fast of 10-12heures . Prior to the intervention, the clinical history including anthropometric measurements and dietary questionnaire (24eures reminder) will be filled out and participants will be asked to rest for 30 min prior to taking their blood pressure at the time of admission, and they should be seated, upright and with their feet on the floor during the process; the measurement will be performed using a manometer on the left arm, elevated at the level of the heart. Afterwards, samples (urine and blood) were taken. Those corresponding to urine will be taken a basal sample (T=0) in a collection bottle. Once the hibiscus-based drink or placebo is ingested, samples will be collected at the following times: 3h, 6h, 12h and 24h. The samples corresponding to blood will be collected with the help of collecting tubes by venous puncture. Eight samples were taken, the first one at the arrival of the patients being basal time (T=B), then at 30 minutes (T=2), 1heure (T=3), 1:30heures (T=4), 2heures (T=5), 3heures (T=6), 4heures (T=7) and 6heures (T=8) after having ingested the hibiscus-based drink or the placebo. During the intervention the volunteers will receive a Western-type diet after the consumption of the beverage, characterized by excessive consumption of red meat, simple carbohydrates, ultra-processed products, colorants, saturated fats, refined sugars and very little intake of fiber and vitamins. After a washout period of more than 6 days, the participants will undergo a second intervention with a different product than the first time (beverage to be evaluated or placebo as appropriate), and the sampling will be repeated.

The second stage will correspond to the evaluation of the glycemic response (GR) and insulinemic response (IR) of the selected individuals. For this purpose, volunteers should come with homogenized dietary conditions (normocaloric and carbohydrate-controlled diet (300 g/day)), without having performed intense physical activity and with a fasting state of 12 hours; In the place they will consume the treatment drink (BT) and the placebo drink (BP) of 60 mL, accompanied by a portion of white bread, so that the sum of the drink plus the white bread will be 50 g of carbohydrates, the administration of the type of drink will be carried out in different sessions, separated by a washout period of 7 days, so that the participants will consume a different one in each session. The RG and RI will be evaluated at time 0 (preprandial), and at 15, 30, 45, 60, 90, and 120 minutes (postprandial), through capillary blood obtained by fingertip puncture. The evaluation corresponding to the GR will be done by taking the second drop and placing it on highly sensitive test strips of the OneTouch Ultra® System, continuing with the determination of the RI through the collection of blood in BD Microtainer SST tubes, which will be centrifuged for 10 minutes (5000 rpm, 25°C) to obtain the serum, which will be used when employing an ELISA human insulin kit.

The study will be carried out at the Nutricia clinic located in Building M of the Instituto Tecnológico y de Estudios Superiores de Occidente (ITESO) located at Anillo Perif. Sur Manuel Gómez Morín 8585, Santa María Tequepexpan, 45604 Tlaquepaque, Jalisco.

ELIGIBILITY:
Inclusion Criteria:

* Normolipidemia Total cholesterol (plasma) < 200 mg/L-1
* Triglycerides < 150 mg/L-1
* Normoglycemia Fasting glucose (plasma) < 100 mg/L-1
* IMC [kg/m2]1 18.5 - 24.9
* Abdominal circumference [cm] Men<90 Women < 80
* Percentage of fat [%] Men<19 Women < 33Systolic pressure [mmHg] < 140
* Diastolic pressure [mmHg] < 90
* Alcohol Last consumption one and a half weeks

Exclusion Criteria:

* Hypertension
* Diabetes
* Smokers
* Cardiovascular disease
* Secondary hyperlipidemia
* Renal insufficiency
* Hyperthyroidism
* In diet
* Pregnant or lactating women, and if their menstrual cycle is close (1 week)
* In medical treatment / supplements
* Hepatic insufficiency
* Infection / inflammatory disease (6 weeks prior to study)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Bioavalability of fenolics compunds and organic acids | the time period will be determined in a single day by evaluating absorption at 0, 0.5, 1, 2, 3, 4, 5 and 6 hours in plasma and for urine its excretion evaluated at 0, 3, 6, 12, 24 hours.
  identification and quantification of bioactive compounds in plasma and urine samples by HPLC-DAD-MS liquid chromatography.
Glycemic response 0 minutes (preprandial) and de next repsponse at 15, 30, 45, 60, 90 and 120 minutes | With the use of this equiment, measurements will be obtained from 0 minutes (preprandial) and at 15, 30, 45, 60, 90 and 120 minutes (postprandial) response
  To obtain the biological sample, a lancet will be used to puncture the pad of the voluntary finger and the sample will be collected in high-sensitivity reactive strips for the measurement of capillary glucose of the OneTouch Ultra System. The portable systeme used for pre- and postprandial glucose measurement allows the monitoring of the capillary glycemic response under experimental conditions for healthy subjects. With the use of this equipment, preprandial and postprandial measurements will be obtained.
Insulinemic response 0 minutes (pre-prandial) | The obtaining of the samples will be taken at 0 minutes (pre-prandial)
  Blood samples will be drawn via capillary puncture. Measurements over time will be similar to the glycemic response assessment techniqeu. Samples will be placed in BD Microtainer SST tubes and kept at room temperature for 30 min. The samples will be centrifucated to obtain serum. Serum insulin concentrations will be analyzed using a solid-phase two-site enzyme immunoassay kit (Human Insulin ElLISA kit, Millipore, EZHI-14K)
Insulinemic response15 minutes | The obtaining of the samples will be taken at 15 minutes
  Blood samples will be drawn via capillary puncture. Measurements over time will be similar to the glycemic response assessment techniqeu. Samples will be placed in BD Microtainer SST tubes and kept at room temperature for 30 min. The samples will be centrifucated to obtain serum. Serum insulin concentrations will be analyzed using a solid-phase two-site enzyme immunoassay kit (Human Insulin ElLISA kit, Millipore, EZHI-14K)
Insulinemic response 30 minutes | The obtaining of the samples will be taken at 30 minutes
  Blood samples will be drawn via capillary puncture. Measurements over time will be similar to the glycemic response assessment techniqeu. Samples will be placed in BD Microtainer SST tubes and kept at room temperature for 30 min. The samples will be centrifucated to obtain serum. Serum insulin concentrations will be analyzed using a solid-phase two-site enzyme immunoassay kit (Human Insulin ElLISA kit, Millipore, EZHI-14K)
Insulinemic response 45minutes | The obtaining of the samples will be taken at 45minutes
  Blood samples will be drawn via capillary puncture. Measurements over time will be similar to the glycemic response assessment techniqeu. Samples will be placed in BD Microtainer SST tubes and kept at room temperature for 30 min. The samples will be centrifucated to obtain serum. Serum insulin concentrations will be analyzed using a solid-phase two-site enzyme immunoassay kit (Human Insulin ElLISA kit, Millipore, EZHI-14K)
markers of inflammation IL-6 | The blood samples will take with the help of collecting tubes by venous puncture, with 8 samples, t=0, then at 30 minutes, 1, 2, 3, 4 5 and 6 hours and Urine samples will be collected at 0, 3,6, 12, 24 hours
  To perform an assay of inflammation markers by proquantum kit specifically interleukin-6 to visualize the decrease of these markers.

SECONDARY OUTCOMES:
Anthropometry measurements | only measure
  measurements will be taken with the Inbody 770 equipment, whose results include weight, height, fat percentages and body muscle mass on the same day to evaluate the volunteers' measurements on the day of the intervention.
Food intake | 2 weeks for the response
  Using Food Frecuency Quertionnaire and 24 hours reminder

CONTACTS AND LOCATIONS:
Locations (1):
- ITESO, Tlaquepaque, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
All information provided by participant is strictly confidential, will be used only by the project's research team and will not be available for any other purpose. The results obtained from this study will be published for scientific purposes but the confidentiality of the participants will never be violated. The information or evidence obtained will be eliminated after fulfilling the scientific purposes for which this intervention was proposed.

REFERENCES:
- [Background] Wolever TM, Jenkins DJ. The use of the glycemic index in predicting the blood glucose response to mixed meals. Am J Clin Nutr. 1986 Jan;43(1):167-72. doi: 10.1093/ajcn/43.1.167. PMID 3942088
- [Background] Sayago-Ayerdi SG, Goni I. [Hibiscus sabdariffa L: source of antioxidant dietary fiber]. Arch Latinoam Nutr. 2010 Mar;60(1):79-84. Spanish. PMID 21090279
- [Background] Marhuenda J, Perez S, Victoria-Montesinos D, Abellan MS, Caturla N, Jones J, Lopez-Roman J. A Randomized, Double-Blind, Placebo Controlled Trial to Determine the Effectiveness a Polyphenolic Extract (Hibiscus sabdariffa and Lippia citriodora) in the Reduction of Body Fat Mass in Healthy Subjects. Foods. 2020 Jan 6;9(1):55. doi: 10.3390/foods9010055. PMID 31935957
- [Background] Hossain MM, Tovar J, Cloetens L, Florido MTS, Petersson K, Prothon F, Nilsson A. Oat Polar Lipids Improve Cardiometabolic-Related Markers after Breakfast and a Subsequent Standardized Lunch: A Randomized Crossover Study in Healthy Young Adults. Nutrients. 2021 Mar 18;13(3):988. doi: 10.3390/nu13030988. PMID 33803802
- [Background] Janson B, Prasomthong J, Malakul W, Boonsong T, Tunsophon S. Hibiscus sabdariffa L. calyx extract prevents the adipogenesis of 3T3-L1 adipocytes, and obesity-related insulin resistance in high-fat diet-induced obese rats. Biomed Pharmacother. 2021 Jun;138:111438. doi: 10.1016/j.biopha.2021.111438. Epub 2021 Mar 13. PMID 33721756
- [Background] Li S, Wu B, Fu W, Reddivari L. The Anti-inflammatory Effects of Dietary Anthocyanins against Ulcerative Colitis. Int J Mol Sci. 2019 May 27;20(10):2588. doi: 10.3390/ijms20102588. PMID 31137777
- [Background] Fernandez-Ochoa A, Cadiz-Gurrea ML, Fernandez-Moreno P, Rojas-Garcia A, Arraez-Roman D, Segura-Carretero A. Recent Analytical Approaches for the Study of Bioavailability and Metabolism of Bioactive Phenolic Compounds. Molecules. 2022 Jan 25;27(3):777. doi: 10.3390/molecules27030777. PMID 35164041
- [Background] Achour M, Bravo L, Sarria B, Ben Fredj M, Nouira M, Mtiraoui A, Saguem S, Mateos R. Bioavailability and nutrikinetics of rosemary tea phenolic compounds in humans. Food Res Int. 2021 Jan;139:109815. doi: 10.1016/j.foodres.2020.109815. Epub 2020 Oct 20. PMID 33509454
- [Background] Sayago-Ayerdi SG, Venema K, Tabernero M, Sarria B, Bravo L, Mateos R. Bioconversion of polyphenols and organic acids by gut microbiota of predigested Hibiscus sabdariffa L. calyces and Agave (A. tequilana Weber) fructans assessed in a dynamic in vitro model (TIM-2) of the human colon. Food Res Int. 2021 May;143:110301. doi: 10.1016/j.foodres.2021.110301. Epub 2021 Mar 10. PMID 33992321

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05774613/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05774613/ICF_001.pdf